CLINICAL TRIAL: NCT02754531
Title: Comparison Between Ultrasonography and Cole Formula in Predicting Uncuffed Endotracheal Tube Diameter
Brief Title: Ultrasonography vs Cole Formula to Predict Endotracheal Tube Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Aida Rosita Tantri SpAn-KA, Consultant, Anesthesiologist, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes006
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: General Anesthesia
Keywords: Cole formula; Pediatric patients; intubation; Ultrasonography; Endotracheal tube; uncuffed; pediatric

ARMS (1):
- Subjects (Experimental): USG was used to measure the internal transversal subglottic diameter on the crichoid cartilago level while the head was in sniffing position. After USG measurement was recorded, Cole formula was used to measure internal diameter of uncuffed endotracheal tube.
  Interventions: Device: USG; Other: Cole Formula

INTERVENTIONS:
Device: USG — USG used was SonoSite® M-Turbo Bothell, WA, USA, probe linear (Array HFL 38 frekuensi 6-13 MHz). Internal subglottic diameter equals external diameter of the uncuffed endotracheal tube or trachea diameter, result rounded to the smallest uncuffed endotracheal tube size.
Other: Cole Formula — Internal diameter of the uncuffed endotracheal tube equals (age in years/4) + 4mm.

SUMMARY:
This study aims to compare the accuracy of measurement between ultrasonography and Cole formula in predicting uncuffed endotracheal tube diameter.

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Non-invasive blood pressure (NIBP) monitor, ECG and pulse-oximeter was set on the subjects in the operation room. The uncuffed endotracheal tube (ETT) diameter predictions were measured firstly using ultrasonography (USG), then with Cole formula. After that, polyvinyl chloride (Mallinckrodt) ETT intubation with Cole diameter measurement was inserted using direct laryngoscopy. If the ETT was too small, use a 0.5 mm bigger ETT than the prediction diameter, if it too big, use a 0.5 mm smaller ETT than the prediction diameter. Reintubation and measurements using both methods were recorded. If bradycardia or desaturation happened, positive pressure ventilation, 100% oxygen, atropine 0,01-0,02 mg/kg, adrenaline 0,01 mg/kg could be given. Data was analyzed using SPSS using Bivariat Chi-square test or Fisher Exact Test (categorical comparative analytical study).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 1-6 years old, Malayan race, planned to undergo elective surgery with general anesthesia with intubation
* Subjects with ASA status I-II
* Cooperative subjects
* Subjects whose parents had signed the informed consent

Exclusion Criteria:

* Subjects with allergies to Ultrasonography jelly
* Subjects with difficult airway
* Subjects with mass in the neck area
* Subjects with respiratory diseases
* Subjects with growth & development disorders
* Subjects with malnutrition (<5% percentile) and obesity (>95% percentile).

Drop out criteria:

* Subjects with cardiorespiratory disorder during intubation
* Subjects who were failed to be intubated twice.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The accuracy proportion of USG and Cole Formula | 3 months
  Whether the USG measurement and Cole Formula measurement accurate or not will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aida R Tantri, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta K, Gupta PK, Rastogi B, Krishan A, Jain M, Garg G. Assessment of the subglottic region by ultrasonography for estimation of appropriate size endotracheal tube: A clinical prospective study. Anesth Essays Res. 2012 Jul-Dec;6(2):157-60. doi: 10.4103/0259-1162.108298. PMID 25885609
- [Background] Park HP, Hwang JW, Lee JH, Nahm FS, Park SH, Oh AY, Jeon YT, Lim YJ. Predicting the appropriate uncuffed endotracheal tube size for children: a radiograph-based formula versus two age-based formulas. J Clin Anesth. 2013 Aug;25(5):384-387. doi: 10.1016/j.jclinane.2013.01.015. Epub 2013 Aug 17. PMID 23965215
- [Background] COLE F. Pediatric formulas for the anesthesiologist. AMA J Dis Child. 1957 Dec;94(6):672-3. doi: 10.1001/archpedi.1957.04030070084009. No abstract available. PMID 13478300
- [Background] Eipe N, Barrowman N, Writer H, Doherty D. A weight-based formula for tracheal tube size in children. Paediatr Anaesth. 2009 Apr;19(4):343-8. doi: 10.1111/j.1460-9592.2008.02916.x. Epub 2009 Jan 21. PMID 19178655
- [Background] van den Berg AA, Mphanza T. Choice of tracheal tube size for children: finger size or age-related formula? Anaesthesia. 1997 Jul;52(7):701-3. doi: 10.1111/j.1365-2044.1997.az0130c.x. PMID 9254579
- [Background] Shibasaki M, Nakajima Y, Ishii S, Shimizu F, Shime N, Sessler DI. Prediction of pediatric endotracheal tube size by ultrasonography. Anesthesiology. 2010 Oct;113(4):819-24. doi: 10.1097/ALN.0b013e3181ef6757. PMID 20808208
- [Background] Bae JY, Byon HJ, Han SS, Kim HS, Kim JT. Usefulness of ultrasound for selecting a correctly sized uncuffed tracheal tube for paediatric patients. Anaesthesia. 2011 Nov;66(11):994-8. doi: 10.1111/j.1365-2044.2011.06900.x. Epub 2011 Sep 20. PMID 21933159
- [Background] Schramm C, Knop J, Jensen K, Plaschke K. Role of ultrasound compared to age-related formulas for uncuffed endotracheal intubation in a pediatric population. Paediatr Anaesth. 2012 Aug;22(8):781-6. doi: 10.1111/j.1460-9592.2012.03889.x. Epub 2012 May 21. PMID 22612446
- [Background] Delilkan AE. Choice of endotracheal tube in the Malaysian paediatric patient--a guide. Singapore Med J. 1973 Mar;14(1):26-8. No abstract available. PMID 4713016
- [Background] Zahedi-Nejad N, Bakhshayesh-Karam M, Kahkoei S, Abbasi-Dezfoully A, Masjedi MR. Normal dimensions of trachea and two main bronchi in the Iranian population. Pol J Radiol. 2011 Oct;76(4):28-31. PMID 22802851
- [Background] Mi W, Zhang C, Wang H, Cao J, Li C, Yang L, Guo F, Wang X, Yang T. Measurement and analysis of the tracheobronchial tree in Chinese population using computed tomography. PLoS One. 2015 Apr 20;10(4):e0123177. doi: 10.1371/journal.pone.0123177. eCollection 2015. PMID 25894917
- [Background] Adewale L. Anatomy and assessment of the pediatric airway. Paediatr Anaesth. 2009 Jul;19 Suppl 1:1-8. doi: 10.1111/j.1460-9592.2009.03012.x. PMID 19572839
- [Background] Prasad A, Yu E, Wong DT, Karkhanis R, Gullane P, Chan VW. Comparison of sonography and computed tomography as imaging tools for assessment of airway structures. J Ultrasound Med. 2011 Jul;30(7):965-72. doi: 10.7863/jum.2011.30.7.965. PMID 21705729
- [Background] Singh M, Chin KJ, Chan VW, Wong DT, Prasad GA, Yu E. Use of sonography for airway assessment: an observational study. J Ultrasound Med. 2010 Jan;29(1):79-85. doi: 10.7863/jum.2010.29.1.79. PMID 20040778
- [Background] Prasanna Kumar S, Ravikumar A. Biometric study of the internal dimensions of subglottis and upper trachea in adult Indian population. Indian J Otolaryngol Head Neck Surg. 2014 Jan;66(Suppl 1):261-6. doi: 10.1007/s12070-012-0477-x. Epub 2012 Jan 21. PMID 24533395
- [Background] CROTEAU JR, COOK CD. Volume-pressure and length-tension measurements in human tracheal and bronchial segments. J Appl Physiol. 1961 Jan;16:170-2. doi: 10.1152/jappl.1961.16.1.170. No abstract available. PMID 13696635
- [Background] Griscom NT, Wohl ME. Dimensions of the growing trachea related to age and gender. AJR Am J Roentgenol. 1986 Feb;146(2):233-7. doi: 10.2214/ajr.146.2.233. PMID 3484568
- See also: Black A, Flynn P, Popat M, Smith H, Thomas M, Wilkinson K. Unanticipated difficult tracheal intubation - during routine induction of anaesthesia in a child aged 1 to 8 years. 2015 — http://www.das.uk.com/